CLINICAL TRIAL: NCT03923335
Title: The Predictive Value of Guangzhou Panel for Recurrence in Early-stage Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: Luo-20190326
Record Dates: First submitted 2019-04-14; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; prognostic biomarkers; DNA Methylation; gene panel; recurrence; disease free survival
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue specimen from colorectal cancer patients who underwent radical resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-risk group: patients with any of the four genes hypermethylated
  Interventions: Other: DNA methylation detection
- low-risk group: patients with none of the four genes hypermethylated
  Interventions: Other: DNA methylation detection

INTERVENTIONS:
Other: DNA methylation detection — detecting the methylation status of colorectal cancer specimen

SUMMARY:
This study aims to evaluate the predictive value of a four-gene methylation assay called Guangzhou Panel in early-stage colorectal cancer. Patients will be divided into two groups: high risk group and low risk group. The primary endpoint is 5 year disease free survival (DFS).

DETAILED DESCRIPTION:
The current risk stratification system defined by clinicopathological features does not identify the risk of disease recurrence in patients with early-stage colorectal cancer (CRC) with optimal accuracy. The investigators aimed to investigate whether the epigenetic alterations could serve as novel prognostic biomarkers that would improve the accuracy of the current primary tumor, regional nodes, metastasis (TNM) staging system.

In the current study, the Investigators have analyzed the genome-wide methylation status of cytosine-phosphate-guanosine (CpG) sites using Infinium MethylationEPIC array in primary tumor and adjacent normal samples from 23 recurrent and 22 recurrence-free stage I and II CRC patients to identify potential methylation markers for disease-free survival (DFS). The prognostic value of the candidate biomarkers has been evaluated in a training cohort (n=174) and an independent validation cohort (n=267), and is to be validated in a prospective cohort (estimated n=287).

Comprehensive data analysis identified a subset of methylated CpG loci that associated with a high risk of recurrence. Methylated CpGs in four genes were significantly associated with DFS in multivariate analysis in both training and validation cohort. Moreover, Hypermethylated Genes Counts panel using these four markers showed a higher prognostic value than any clinicopathological factor, current molecular biomarkers or single methylated CpG marker alone in the training and validation cohorts. This four-gene methylation assay is defined as Guangzhou Panel.

The investigators aim to conduct a prospective observational study to evaluate the predictive value of Guangzhou Panel in early-stage colorectal cancer. A total of 287 patients with pathologically verified stage I-II CRC and underwent surgical resection are expected to be recruited in our study. These patients will be divided into high-risk group and low-risk group and will be followed up at least 5 years. The primary endpoint is 5-year disease free survival (DFS). The prognostic strength of candidate biomarkers was adjusted in multivariate Cox regression models including multiple biomarkers and clinicopathologic variables.

ELIGIBILITY:
Inclusion Criteria:

1. TNM stage I-II (T1-4N0M0) colorectal cancer cases
2. receive radical surgical resection
3. have completed data of tumor location, histological type, behavioral characteristics or TNM staging
4. have tumor specimens and either a valid microsatellite instability (MSI) or immuno-histochemistry (IHC) data
5. have valid V-raf murine sarcoma viral oncogene homolog B1 (BRAF), kirsten rat sarcoma viral oncogene (KRAS), CpG island methylator phenotype (CIMP) results
6. have at least 4 years of follow-up
7. have valid time to local recurrence/metastasis in follow-up
8. have clinical/treatment record data and valid preoperative status of intestinal obstruction or perforation (IOP), counts of lymph node removed in surgical resection.

Exclusion Criteria:

1. have had a previous diagnosis of any cancer or presence of any tumor other than the CRC
2. have had inflammatory bowel disease
3. have had hereditary colorectal cancer syndromes, including Familial adenomatous polyposis, mutyh (MYH)-associated polyposis, Peutz-Jeghers syndrome, Juvenile polyposis coli, phosphate and tension homology deleted on chromosome ten (PTEN) tumor-hamartoma syndromes, Lynch Syndrome, and Familial Colorectal Cancer Type X.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that had pathologically verified stage I-II CRC and underwent surgical resection in Sixth Affiliate Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 287 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | From date of operation until the date of first recurrence or date of death from any cause, whichever came first, assessed up to 5 years
  the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yanxin Luo, MD,PhD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Our DNA methylation panel is applying for patent protection, therefore we plan to keep the data private for the time being.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] O'Connor ES, Greenblatt DY, LoConte NK, Gangnon RE, Liou JI, Heise CP, Smith MA. Adjuvant chemotherapy for stage II colon cancer with poor prognostic features. J Clin Oncol. 2011 Sep 1;29(25):3381-8. doi: 10.1200/JCO.2010.34.3426. Epub 2011 Jul 25. PMID 21788561
- [Background] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Background] Quasar Collaborative Group; Gray R, Barnwell J, McConkey C, Hills RK, Williams NS, Kerr DJ. Adjuvant chemotherapy versus observation in patients with colorectal cancer: a randomised study. Lancet. 2007 Dec 15;370(9604):2020-9. doi: 10.1016/S0140-6736(07)61866-2. PMID 18083404
- [Background] Morris EJ, Maughan NJ, Forman D, Quirke P. Who to treat with adjuvant therapy in Dukes B/stage II colorectal cancer? The need for high quality pathology. Gut. 2007 Oct;56(10):1419-25. doi: 10.1136/gut.2006.116830. Epub 2007 May 9. PMID 17494107
- [Background] Ribic CM, Sargent DJ, Moore MJ, Thibodeau SN, French AJ, Goldberg RM, Hamilton SR, Laurent-Puig P, Gryfe R, Shepherd LE, Tu D, Redston M, Gallinger S. Tumor microsatellite-instability status as a predictor of benefit from fluorouracil-based adjuvant chemotherapy for colon cancer. N Engl J Med. 2003 Jul 17;349(3):247-57. doi: 10.1056/NEJMoa022289. PMID 12867608
- [Background] Kennedy RD, Bylesjo M, Kerr P, Davison T, Black JM, Kay EW, Holt RJ, Proutski V, Ahdesmaki M, Farztdinov V, Goffard N, Hey P, McDyer F, Mulligan K, Mussen J, O'Brien E, Oliver G, Walker SM, Mulligan JM, Wilson C, Winter A, O'Donoghue D, Mulcahy H, O'Sullivan J, Sheahan K, Hyland J, Dhir R, Bathe OF, Winqvist O, Manne U, Shanmugam C, Ramaswamy S, Leon EJ, Smith WI Jr, McDermott U, Wilson RH, Longley D, Marshall J, Cummins R, Sargent DJ, Johnston PG, Harkin DP. Development and independent validation of a prognostic assay for stage II colon cancer using formalin-fixed paraffin-embedded tissue. J Clin Oncol. 2011 Dec 10;29(35):4620-6. doi: 10.1200/JCO.2011.35.4498. Epub 2011 Nov 7. PMID 22067406
- [Background] Esteller M. Epigenetics in cancer. N Engl J Med. 2008 Mar 13;358(11):1148-59. doi: 10.1056/NEJMra072067. No abstract available. PMID 18337604
- [Background] Feinberg AP. The Key Role of Epigenetics in Human Disease Prevention and Mitigation. N Engl J Med. 2018 Apr 5;378(14):1323-1334. doi: 10.1056/NEJMra1402513. No abstract available. PMID 29617578
- [Background] Weisenberger DJ, Siegmund KD, Campan M, Young J, Long TI, Faasse MA, Kang GH, Widschwendter M, Weener D, Buchanan D, Koh H, Simms L, Barker M, Leggett B, Levine J, Kim M, French AJ, Thibodeau SN, Jass J, Haile R, Laird PW. CpG island methylator phenotype underlies sporadic microsatellite instability and is tightly associated with BRAF mutation in colorectal cancer. Nat Genet. 2006 Jul;38(7):787-93. doi: 10.1038/ng1834. Epub 2006 Jun 25. PMID 16804544
- [Background] Brock MV, Hooker CM, Ota-Machida E, Han Y, Guo M, Ames S, Glockner S, Piantadosi S, Gabrielson E, Pridham G, Pelosky K, Belinsky SA, Yang SC, Baylin SB, Herman JG. DNA methylation markers and early recurrence in stage I lung cancer. N Engl J Med. 2008 Mar 13;358(11):1118-28. doi: 10.1056/NEJMoa0706550. PMID 18337602
- [Background] Hinoue T, Weisenberger DJ, Lange CP, Shen H, Byun HM, Van Den Berg D, Malik S, Pan F, Noushmehr H, van Dijk CM, Tollenaar RA, Laird PW. Genome-scale analysis of aberrant DNA methylation in colorectal cancer. Genome Res. 2012 Feb;22(2):271-82. doi: 10.1101/gr.117523.110. Epub 2011 Jun 9. PMID 21659424
- [Background] Luo Y, Wong CJ, Kaz AM, Dzieciatkowski S, Carter KT, Morris SM, Wang J, Willis JE, Makar KW, Ulrich CM, Lutterbaugh JD, Shrubsole MJ, Zheng W, Markowitz SD, Grady WM. Differences in DNA methylation signatures reveal multiple pathways of progression from adenoma to colorectal cancer. Gastroenterology. 2014 Aug;147(2):418-29.e8. doi: 10.1053/j.gastro.2014.04.039. Epub 2014 Apr 30. PMID 24793120
- [Background] Martinez-Cardus A, Moran S, Musulen E, Moutinho C, Manzano JL, Martinez-Balibrea E, Tierno M, Elez E, Landolfi S, Lorden P, Arribas C, Muller F, Bock C, Tabernero J, Esteller M. Epigenetic Homogeneity Within Colorectal Tumors Predicts Shorter Relapse-Free and Overall Survival Times for Patients With Locoregional Cancer. Gastroenterology. 2016 Nov;151(5):961-972. doi: 10.1053/j.gastro.2016.08.001. Epub 2016 Aug 10. PMID 27521480
- [Background] Pidsley R, Zotenko E, Peters TJ, Lawrence MG, Risbridger GP, Molloy P, Van Djik S, Muhlhausler B, Stirzaker C, Clark SJ. Critical evaluation of the Illumina MethylationEPIC BeadChip microarray for whole-genome DNA methylation profiling. Genome Biol. 2016 Oct 7;17(1):208. doi: 10.1186/s13059-016-1066-1. PMID 27717381
- [Background] Moran S, Arribas C, Esteller M. Validation of a DNA methylation microarray for 850,000 CpG sites of the human genome enriched in enhancer sequences. Epigenomics. 2016 Mar;8(3):389-99. doi: 10.2217/epi.15.114. Epub 2015 Dec 17. PMID 26673039